CLINICAL TRIAL: NCT00999440
Title: QTc and Perceived Sleep Follow up Among Chronic Pain Patients With Opiate Medication
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Tel-Aviv Sourasky Medical Center, Pain Medicine Unit, Tel-Aviv Sourasky Medical Center, Pain Medicine Unit
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMC-09-SB-0104-09-CTIL
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2010-01-21 (Estimated); Status verified 2009-12

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; Methadone; Perceived Sleep; QTc
MeSH Terms: conditions — Chronic Pain | interventions — Methadone

ARMS (1):
- Methadone (Experimental): ECG (QT, QTc, Heart rate), Urine sample (opiates, benzodiazepines, THC, cocaine, amphetamines, methadone-metabolite), Questionnaire PSQI - perceived sleep - self report , Pain indices (severity, duration, cause, etc.) , usage of other medication for pain and other significant disease/disorders, history of drug abuse, age, sex, place of birth and ethnic origin, comorbidity. Follow up after 4weeks, 6months and 1 year will be done.Patients who start with any opiate and then switch to methadone, move to methadone follow up
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Methadone — ECG (QT, QTc, Heart rate), Urine sample (opiates, benzodiazepines, THC, cocaine, amphetamines, methadone-metabolite), Questionnaire PSQI - perceived sleep - self report , Pain indices (severity, duration, cause, etc.) , usage of other medication for pain and other significant disease/disorders, history of drug abuse, age, sex, place of birth and ethnic origin, comorbidity. Follow up after 4weeks, 6months and 1 year will be done. Patients who start with any opiate and then switch to methadone, move to methadone follow up

SUMMARY:
QTc:

Since the reports of three deaths attributed to Torsade de Point (TdP) related to treatment with the long-acting methadone derivative levomethadyl acetate HCl (LAAM), methadone has been scrutinized for any possible association with TdP. Since then, several studies among Methadone Maintenance Treatment (MMT) patients and chronic pain patients were done, reporting diverse results about possible association between methadone dose and QTc prolongation. Most studies however were cross-sectional and generally found insignificant clinical prolongation of QTc. A follow up studies are of importance, and although few studies have started evaluating QTc among MMT patients, none was done among chronic pain patients with no history of drug usage. One study of 8 chronic pain patients experiencing insufficient pain control or intolerable side effects during treatment with oral morphine switched to oral methadone showed insignificant modest increase QTc following 9 month.

Perceived Sleep:

Chronic pain patients as well as drug addicts are known to suffer from poor sleep. Some studies found possible relation to methadone dose, however, no causal association was found and importantly some also found association with duration of opiate usage before starting methadone when entry to MMT clinic. Thus, patients with no history of opiate addiction are an important interesting group that may help understand relation between methadone usage and sleep quality. However, sleep must be evaluate before opiate administration and a follow up study is needed

ELIGIBILITY:
Inclusion Criteria:

* adults (18+ years) patients with chronic pain, who intend to be medicated with any opiates

Exclusion Criteria:

* patient with no opiate usage through last year

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the influence of opioid drugs on QTc interval before and during Opioid treatment among patients suffering from chronic pain. | 1 year

SECONDARY OUTCOMES:
To evaluate the perceived sleep in the chronic pain patients | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Pain Medicine Unit, Tel Aviv, Israel